CLINICAL TRIAL: NCT00271973
Title: The Pharmacogenetics of Oxycodone Analgesia in Human Experimental Pain Models
Brief Title: OXY-2: The Pharmacogenetics of Oxycodone Analgesia in Human Experimental Pain Models
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EudraCT 2005-004082-42
Record Dates: First submitted 2006-01-03; First posted 2006-01-04 (Estimated); Last update posted 2007-01-30 (Estimated); Status verified 2007-01

CONDITIONS: Healthy
MeSH Terms: interventions — Oxycodone

INTERVENTIONS:
Drug: Oxycodone

SUMMARY:
Thirty-two healthy volunteers will be submitted to experimental pain and on the 2 study days receive Oxycodone 20 mg po vs. placebo. Half of the volunteers will be poor metabolizers according to CYP2D6 genotype and half will be extensive metabolizers (EM) and have an enzyme with normal function. The study hypothesis is that PM will experience less pain relief than EM.

DETAILED DESCRIPTION:
Oxycodone is a semi-synthetic opioid with an analgesic effect in the postoperative pain management comparable to morphine. Oxycodone is N-demethylated by CYP2D6 to its active metabolite oxymorphone, a potent μ-receptor agonist. A genetic polymorphism divides a Caucasian population into two groups: 8% with an enzyme lacking activity, poor metabolizers (PM) and the rest with normal CYP2D6 activity, extensive metabolizers (EM).

Many different, single nucleotide polymorphisms (SNPs) are responsible for interindividual differences in the effect of opioids. Among these are the A118G SNP in the μ-receptor gene OPRM1 and the C3435T and G2677T/A SNPs in the MDR-1 gene of P-glycoprotein. P-glycoprotein is responsible for the absorption, excretion and transport of many drugs including opioids over the blood-brain barrier.

Electrical stimulation and cold pressor test are among the most well defined and evaluated human experimental pain models. The 32 volunteers will be submitted to the tests before and 1, 2, 3 and 4 hours after medicine intake.

To determine the plasma levels of Oxycodone and its metabolites blood will be drawn after each pain test. Also the CYP2D6 genotype and the above mentioned SNPs will be determined from the blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer age between 20 and 40 years.
* Healthy according to medical history and physical examination.
* Informed consent given.
* Phenotyped or genotyped as extensive or poor metabolizer of sparteine.
* Female: Use of safe contraception (IUD, gestagen injectiones or oral contraceptive) or negative u-HCG test.

Exclusion Criteria:

* Any known allergy or intolerance to oxycodone.
* Regularly drug therapy or medication (except contraceptives).
* Alcohol or medicine abuse.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32
Dates: Start 2006-02; Study Completion 2007-01

PRIMARY OUTCOMES:
Pain threshold and tolerance measured by electrical stimulation and pain intensity measured by cold pressor test.

SECONDARY OUTCOMES:
The above compared to SNPs. Plasma levels of oxycodone and metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: Stine T. Zwisler, Dr., Principal Investigator — University of Southern Denmark
Locations (1):
- University of Southern Denmark, IST Clinical Pharmacology, Odense, Odense C, Denmark